CLINICAL TRIAL: NCT00673166
Title: Evaluation of Local Mechanisms for Staff Motivation to Improve Treatment and Reduce Mortality Due to Malaria at the Paediatric Ward
Brief Title: Evaluation of Local Mechanisms for Staff Motivation to Reduce Hospital Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HMTV; GMP_P_II_5
Record Dates: First submitted 2008-05-01; First posted 2008-05-07 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Hospital Mortality; Malaria
Keywords: Staff motivation; Hospital mortality; Perception of quality of care
MeSH Terms: conditions — Malaria | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Staff incentive & supervision — Control & management of funds for incentive of staff; supervision
Behavioral: Staff motivation — Supervision, control of funds

SUMMARY:
We observed in a randomised intervention trial in Bissau that mortality due to malaria could be reduced by half by adding a small monetary incentive to the staff and strict follow-up of a standard protocol for available drugs. The Government and donors are not able to sustain such incentives. We intend to evaluate whether strict organisation of a cost recovery system and the use of part of the funds for staff incentives would improve performance of the staff and contribute to reduction of hospital and post-discharge mortality.

DETAILED DESCRIPTION:
A committee will organise collection and use of the money, and decide on incentives to be paid to the staff based on performance indicators. All children < 5 years of age admitted to the ward will be registered and followed-up until two months after the consultation. Data on the level of mortality before and after the study period will be collected. Furthermore, interviews on quality perception of the parents will be carried out before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* Children under five years of age admitted to the ward
* Parents of these children

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall hospital and malaria mortality | One year

SECONDARY OUTCOMES:
Parent's perception of the quality of care received | One year

CONTACTS AND LOCATIONS:
Overall Officials: Amabelia Rodrigues, PhD, Principal Investigator — Bandim Health Project & Gates Malaria Partnership
Locations (1):
- Paediatric department at the national hospital, Bissau, Bissau Region, Guinea-Bissau

REFERENCES:
- [Background] Biai S, Rodrigues A, Gomes M, Ribeiro I, Sodemann M, Alves F, Aaby P. Reduced in-hospital mortality after improved management of children under 5 years admitted to hospital with malaria: randomised trial. BMJ. 2007 Oct 27;335(7625):862. doi: 10.1136/bmj.39345.467813.80. Epub 2007 Oct 22. PMID 17954513
- [Background] Sodemann M, Veirum J, Biai S, Nielsen J, Bale C, Skytte Jakobsen M, Gustafson P, Aaby P. Reduced case fatality among hospitalized children during a war in Guinea-Bissau: a lesson in equity. Acta Paediatr. 2004 Jul;93(7):959-64. PMID 15303813